CLINICAL TRIAL: NCT05544266
Title: Rare and Atypical Diabetes Network
Acronym: RADIANT
Status: Recruiting | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: RADIANT; 5U54DK118638 (NIH); 5U54DK118612 (NIH)
Record Dates: First submitted 2022-08-23; First posted 2022-09-16 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus Progression; Glucose Intolerance; Glucose Metabolism Disorders; Metabolic Disease; Endocrine; Complications; Endocrine System Diseases
Keywords: RADIANT; Atypical Diabetes; Rare Diabetes; Glucose Intolerance
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood Serum Plasma DNA RNA Urine Peripheral Blood Monocytes (PBMCs)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
RADIANT is a network of 14 clinical sites and several laboratories dedicated to the study of atypical diabetes.

The objective of this study is to define new forms of diabetes and the unique mechanisms underlying these forms of atypical diabetes. The specific aims are to:

1. Identify and enroll individuals and families with undiagnosed rare and atypical forms of diabetes.
2. Determine the etiologic basis of the metabolic disorder among individuals and families with novel forms of rare and atypical diabetes.
3. Understand the pathophysiology of individuals and families with novel forms of rare and atypical forms of diabetes.

DETAILED DESCRIPTION:
RADIANT has three distinct stages.

Stage 1:

Stage 1 participants will complete a consent form and a questionnaire to determine the potential for having atypical forms of diabetes. Participants identified as potentially atypical based on questionnaire responses will be asked to provide a blood sample to test for islet autoantibodies and complete additional questionnaires.

The RADIANT Adjudication Committee, which is comprised of a team of experts in diabetes, will assess the data collected in Stage 1 and select and prioritize participants to proceed to Stage 2 and 3 for Whole Genome Sequencing (WGS) and other testing.

Stage 2:

Stage 2 of the study includes genetic screening for known forms of monogenic diabetes. Participants will consent for this stage of the study, complete a family history questionnaire, and have blood collected for DNA and RNA extraction, storage, and analysis. WGS will be performed on all DNA samples. If no pathogenic/likely pathogenic variant in a known monogenic diabetes gene that is thought to explain the participant's diabetes is identified by WGS, RNA Sequencing will be performed at Baylor College of Medicine.

Stage 3:

Stage 3 of the study includes deeper phenotyping. All participants who proceed to Stage 3 will visit a study clinic to consent and complete Stage 3 Standard procedures which include: an Oral Glucose Tolerance Test (OGTT), additional blood collection, a detailed physical exam, and additional questionnaires.

Discovery Team Review:

The work of the Discovery Team is expected to be an iterative process analyzing all data collected up to this point in the study to understand the significance of novel variants. In some instances, the Discovery Team may determine that enrollment of the Proband's family members is necessary. Family members with suspected atypical diabetes will follow the same study procedures as described above. Affected and unaffected family members may also be enrolled for Sanger Sequencing. The Discovery Team may also recommend additional optional procedures to better characterize the participant's form of diabetes.

ELIGIBILITY:
Inclusion Criteria:

The following criteria or phenotypes will be considered for suspecting "atypical" participants:

* Type 2 diabetes diagnosed at a time when the individual was prepubertal or non-obese
* Mendelian pattern, especially with early onset (<18 years old)
* Syndromic (multiple systems involved)
* Lipodystrophic
* Extremes of BMI
* "Mitochondrial" characteristics (e.g., myopathy, hearing deficits)
* Non-progressive
* Rapidly progressive ("fulminant")
* Low insulin requirements (<0.5 u/kg/day)
* Cyclical hyperglycemia with periods of remission
* Lean persons with polycystic ovarian syndrome (PCOS)
* History of gestational diabetes (GDM) when lean
* Lean insulin-resistant persons
* If islet autoantibodies and beta-cell function parameters have been measured (where "A" = islet cell autoantibodies, "B" = beta-cell function):

oA-B- (i.e., lacking islet autoimmunity makers and lacking beta cell function) oA-B+ with unprovoked DKA at initial presentation (i.e., lacking islet autoimmune markers, with preserved beta-cell function, but presenting with unprovoked DKA) oA-B+ of very young onset (pre-pubertal) (i.e., lacking islet autoimmune markers, with preserved beta-cell function, but very early onset T2D-like phenotype)

Exclusion Criteria:

* Those with high likelihood of typical type 1, typical type 2, known monogenic, or other known secondary forms of diabetes
* Refusal of consent for genetic testing
* Islet autoantibody positive (participants who are islet autoantibody positive but present with additional atypical features i.e. syndromic, strong linear family history of diabetes may not be excluded)
* Women who are currently pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Probands and family members will be screened for evaluation of suspected atypical diabetes of unknown origin. Among the pool of evaluated individuals, those found to have a known form of diabetes will be excluded from further study. The remaining participants will be prioritized for genetic/genomic analysis and further testing.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Phenotypic and genotypic characterization of previously unknown forms of diabetes using Whole Genome Sequencing (WGS), and deeper phenotyping methods | Through study completion, an average of 3 years.
  Deeper phenotyping methods include both clinical and laboratory assessments. Clinical data includes anthropometric and biometric data, medical histories, and standard questionnaires (ASA24, PROMIS, environmental exposures depression and anxiety). Laboratory data includes WGS, transcriptomics, metabolomics, mitochondrial sequencing, Oral Glucose Tolerance Test (OGTT), and Islet autoantibodies. Clustering methods will be used to define cohorts of similar diabetes genotypes and phenotypes based on this data.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Krischer, PhD, Study Chair — University of South Florida
Locations (13):
- United States (13):
  - University of Colorado- Denver, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - SUNY Downstate Health Sciences University, Brooklyn, New York
  - Columbia University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] RADIANT Study Group. The Rare and Atypical Diabetes Network (RADIANT) Study: Design and Early Results. Diabetes Care. 2023 Jun 1;46(6):1265-1270. doi: 10.2337/dc22-2440. PMID 37104866